CLINICAL TRIAL: NCT03135158
Title: The Association Between Shock Index and Severity of Postpartum Blood Loss: An Observational Study
Brief Title: The Association Between Shock Index and Severity of Postpartum Blood Loss
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Collaborators: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Sponsor
Other Study IDs: 3009
Record Dates: First submitted 2017-04-20; First posted 2017-05-01 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women in labor: All participants who have a vaginal delivery
  Interventions: Other: Exposure to vaginal delivery

INTERVENTIONS:
Other: Exposure to vaginal delivery — Women who have vaginal births are observed for a minimum of 1 hour postpartum

SUMMARY:
The present study aims to determine the relationship between postpartum changes in the shock index and the severity of blood loss and other PPH results. Blood loss, heart rate and blood pressure will be systematically measured in the postpartum period in all participating women to explore new clinical indicators to identify those requiring clinical intervention for excessive bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Receive care for vaginal delivery

Exclusion Criteria:

* Scheduled or transferred for cesarean section
* Cannot give informed consent
* Are not willing and/or cannot answer the questionnaire on their background

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All women presenting for vaginal delivery will be invited to participate
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Correlation between blood loss and shock index | Within 1 hour postpartum
  Correlate shock index, heart rate, and blood pressure measurements with blood loss levels at 15, 30, 45 & 60 minutes

SECONDARY OUTCOMES:
Percentage of women with blood loss ≥ 500 ml and ≥ 1000 ml | Up to two hours postpartum
  Proportions with ≥ 500 ml and ≥ 1000 ml blood loss at 30 and 60 minutes postpartum, at PPH diagnosis (if applicable), and when active bleeding stops
Median blood loss in the postpartum and interquartile range | Up to two hours postpartum
  Blood loss at 30 and 60 minutes postpartum, at PPH diagnosis (if applicable), and when active bleeding stops
Percentage of women who received treatment to control bleeding | Up to two hours postpartum
Average change in Hb measured before and after delivery | Pre-delivery and at least 24 hours postpartum
  Among women receiving treatment to control postpartum hemorrhage
Percentage of women with complications | Through study completion, an average of 24-48 hours postpartum
  Among women receiving treatment to control postpartum hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Jill Durocher, Principal Investigator — Gynuity Health Projects; Ilana Dzuba, MPH, Principal Investigator — Gynuity Health Projects
Locations (1):
- Fundación Valle del Lili, Cali, Colombia